CLINICAL TRIAL: NCT05986903
Title: Influence of HLA-DQA1*05 Genotype in Adults With Inflammatory Bowel Disease and Anti-TNF Treatment With Proactive Therapeutic Drug Monitoring. A Prospective Multicenter Study.
Brief Title: Influence of HLA-DQA1*05 Genotype in Adults With Anti-TNF Treatment With Proactive Therapeutic Drug Monitoring.
Acronym: Proa-DQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital del Rio Hortega (Other)
Collaborators: Francisco Javier Garcia Alonso (Unknown); Jesús Barrio (Unknown)
Responsible Party: Principal Investigator, Esteban Fuentes-Valenzuela, MD, Hospital del Rio Hortega
Other Study IDs: 22-EO033
Record Dates: First submitted 2023-05-01; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Drug Monitoring; Inflammatory Bowel Diseases
Keywords: proactive therapeutic drug monitoring; HLA-DQA1*05 genotype; Anti-TNF
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Tumor Necrosis Factor-alpha

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HLA-DQA1*05 variant carriers
  Interventions: Drug: Tumor necrosis factor (TNF)-alpha inhibitors
- HLA-DQA1*05 non-carriers
  Interventions: Drug: Tumor necrosis factor (TNF)-alpha inhibitors

INTERVENTIONS:
Drug: Tumor necrosis factor (TNF)-alpha inhibitors — Proactive drug monitoring was defined as the assessment of trough concentrations to optimize dosing during induction therapy and intermittently thereafter regardless of symptoms or inflammatory markers.
  During induction, the following target concentrations are employed: 25-30 mcg/ml (week 2) and 20 mcg/ml (week 6) for Infliximab and > 10 mcg/ml (week 2 and 4) for Adalimumab. Checks are performed systematically at week 2 and 6 (infliximab) and at week 4 (adalimumab).
  During the maintenance, the targets are 5-10 mcg/ml for Infliximab and 8-12 mcg/ml for Adalimumab. In case of perianal disease, the targets are 7-20 mcg/ml.

SUMMARY:
HLA-DQA1*05 variant carriers are at risk of developing antibodies against infliximab and adalimumab with reduced TNF antagonist persistence.

The impact of proactive therapeutic drug monitoring (PTDM) on this association has been barely assessed.

Therefor, we propose a cohort study including adult patients with Crohn's disease and ulcerative colitis treated with TNF antagonists under proactive therapeutic drug monitoring.

Our hypothesis is that, proactive therapeutic drug monitoring could be an alternative to combination treatment with immunomodulators to increase TNF-antagonists' persistence in HLA-DQA1*05 carriers.

DETAILED DESCRIPTION:
Population study: patients with inflammatory bowel disease and initiation of anti-TNF therapy

Inclusion and exclusion criteria

The inclusion criteria are:

* Patient diagnosed with inflammatory bowel disease based on clinical, endoscopic, and pathological criteria according to ECCO criteria.
* Initiation of anti-TNf, including infliximab and adalimumab.
* Subjects naïve to biological treatment
* Age >18 years.

The exclusion criteria are:

* No determination of HLA DQA1*5 allele.
* No proactive drug monitoring
* Initiation of anti-TNF treatment as prevention of post-surgical recurrence in Crohn's disease during the first 12 months after surgery or, after that time, with a colonoscopy with a Rutgeerts 0-1
* Anti-TNF treatment with combined treatment with immunomodulator. Prior initiation of immunomodulator or prior use and suspension would not be a contraindication
* Initiation of anti-TNF treatment for extraintestinal manifestation
* Initiation of anti-TNF treatment during pregnancy.

Proactive drug monitoring was defined as standardized determination of drug levels during induction and maintenance, with optimization independently of the patient's clinical status, until reaching target levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of inflammatory bowel disease according to ECCO criteria.
* Older than 18 years
* Subjects naïve to biological treatment
* Anti-TNF treatment initiation (infliximab or adalimumab) due to intestinal activity and/or perianal disease.
* Avaibility to evaluate HLA DQA1*05 status
* Proactive therapeutic drug monitoring of anti-TNF levels

Exclusion Criteria:

* Initiation of anti-TNF treatment as prevention of post-surgical recurrence in Crohn's disease during the first 12 months after surgery or, afterwards, if endoscopic recurrence with a Rutgeerts 0-1.
* Initiation of anti-TNF treatment under combo treatment with immunomodulator. Prior initiation of immunomodulator or prior use and suspension would not be a contraindication.
* Initiation of anti-TNF treatment due to extraintestinal activity.
* Initiation of anti-TNF treatment by a non-gastroenterologist specialist.
* Initiation of anti-TNF treatment during pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of inflammatory bowel disease (Crohn's disease, ulcerative colitis and indeterminate colitis), who require starting anti-TNF for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Corticosteroid-free clinical remission and treatment maintenance at week 54 | Week 54
  Corticosteroid-free clinical remission was defined as Harvey Bradshaw score <5 for Crohn's disease or partial Mayo score ≤2 for ulcerative colitis with no item exceeding one point, without corticosteroid

SECONDARY OUTCOMES:
Corticosteroid-free clinical response and remission at week 12. | week 12
  Corticosteroid-free clinical response was defined as Harvey Bradshaw score < 5 or a decrease ≥ 3 points from baseline in Crohn's disease. For ulcerative colitis, a decrease in the partial Mayo Index of at least 3 points or 30% accompanied by a decrease in rectal bleeding by one point, without corticosteroid
Proportions of patients with ultrasound remission at week 12 and 24 | week 12 and 24
  Ultrasound remission was defined as SUS-CD 0 for Crohn's disease or a bowel wall thickness < 2.1 mm for ulcerative colitis
Proportions of patients with clinical-biochemical remission at week 54. | week 54
  Clinical-biochemical remission was defined as CRP ≤ 5 mg/L and fecal calprotectin < 150 mg/kg
Proportions of endoscopic remission at week 54 between both groups. | week 54
  For Crohn's disease endoscopic remission was defined as a SES-CD <3 points or absence of ulcerations (e.g. SES-CD ulceration subscores ¼ 0) For ulcerative colitis, a Mayo endoscopic subscore of 0 points, or UCEIS ≤1 points
Proportions of primary failure between both groups | week 12
To compare drug levels at week 6 (infliximab) and week 4 (adalimumab) in subjects with a standard induction | week 4 or 6
  Drug monitoring at week 6 for infliximab and week 4 for adalimumab.
Proportion of subjects with anti-drug antibodies at the end of induction and week 54. | week 54
  Anti-infliximab and anti-adalimumab antibodies at week 4 for adalimumab, at week 6 for infliximab and at week 54 for both.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Rio Hortega, Valladolid, Spain